CLINICAL TRIAL: NCT02212652
Title: The Effect of VItamin D Supplementation on Nutritional STatus and Adverse Outcomes in Bariatric Surgery (VISTA)
Brief Title: Vitamin D to Improve Nutrition Prior to Bariatric Surgery and Investigate the Relationship With Negative Outcomes
Acronym: VISTA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of support resources to complete study appropriately
Sponsor: Johns Hopkins University (Other)
Collaborators: Bariatric Advantage (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00044789
Record Dates: First submitted 2014-08-06; First posted 2014-08-08 (Estimated); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Vitamin D Deficiency; Vitamin D Insufficiency
Keywords: Bariatric surgery; Vitamin D deficiency; Vitamin D insufficiency; Adverse surgical outcomes; Clinical outcomes
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Vitamin D; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care plus Vitamin D (Active Comparator): If randomized to this arm, each participant will receive a 30 day supply of 10,000 IU of VitD3 for research purposes in addition to receiving standard of care. We will ask that they take one of these supplements daily with their largest meal of the day until their surgery.
  Interventions: Dietary Supplement: Vitamin D; Other: Standard of Care
- Standard of Care plus Placebo (Placebo Comparator): If randomized to this arm, each participant will receive a 30 day supply of placebo supplements for research purposes in addition to receiving standard of care. We will ask that they take one of these supplements daily with their largest meal of the day until their surgery.
  Interventions: Other: Placebo; Other: Standard of Care

INTERVENTIONS:
Dietary Supplement: Vitamin D — 10,000 IU of VitD3 daily (one gel daily)
  Other Names: Bariatric Advantage Vitamin D Chewable Gels
  Arms: Standard of Care plus Vitamin D
Other: Placebo — Gummy button placebo, which will appear very similar to the vitamin D supplement.
  Arms: Standard of Care plus Placebo
Other: Standard of Care — Patients will receive the standard care provided to all patients undergoing bariatric surgery regardless of research study participation status.

SUMMARY:
VISTA is looking to see if vitamin D supplements before bariatric surgery might improve vitamin D stores, which may help to prevent some complications like infections.

Who can join this research study?

* Approved to undergo bariatric surgery-Roux-en-Y Gastric Bypass or Vertical Sleeve Gastrectomy-at the Johns Hopkins Bayview Medical Center
* 18 to 64 years of age
* BMI of 35 to 49.9 kg/m2
* VitD insufficient or deficient prior to having surgery

What will happen if a participant chooses to participate in this research study?

* The participant will be randomly assigned (by chance) to receive either:
* Standard care plus vitamin D supplements or
* Standard care plus a placebo (contains no vitamin D)
* Either would be provided at no cost to the participant
* The investigators will ask the participant to complete a survey on the day of surgery regarding supplement use
* The investigators will follow the participants medical record through the 12 month follow up clinic visit.

DETAILED DESCRIPTION:
An estimated 2 in 3 American adults are either overweight (BMI 25-29.9 kg/m2) or obese (BMI 30-39.9 kg/m2). The prevalence of obesity, morbid obesity (BMI 40-44.9 kg/m2), and even super obesity (BMI ≥ 45 kg/m2) are increasing. Obesity is a leading contributor to global mortality and contributes to the burden of disease associated with diabetes, cardiovascular disease, musculoskeletal disorders such as osteoarthritis, and some cancers. Morbid obesity reduces life expectancy by 8 to 10 years, similar to the effect of being a regular cigarette smoker.

Several studies have demonstrated that most obese adults are vitamin D (VitD) insufficient (<75 nmol/L, 30 ng/ml) or deficient (<50 nmol/L, 20 ng/ml). The inverse relationship between body mass index (BMI) or body fat mass and VitD status is hypothesized to be due to sequestration of VitD by adipose tissue, reducing the bioavailability of VitD. The classical role of VitD is in the maintenance of bone calcification, but more recent research has elucidated a more varied role for this hormone. Lack of VitD has been associated with increased susceptibility to infection, autoimmunity, cancer, and chronic disease.

Bariatric surgery is currently the most successful means of long-term weight loss. Since deficiency in fat-soluble vitamins, such as VitD, is considered a metabolic complication of bariatric surgery, determining the VitD status of these individuals and perhaps correcting it prior to surgery may prove greatly beneficial. Potential complications relating to VitD insufficiency and deficiency include adverse surgical outcomes such as improper wound healing, infection of the surgical incision, and atrial fibrillation. Since the indications for bariatric surgery are obesity and obesity-related comorbidities, bariatric surgery patients are at an increased risk of having an adverse surgical outcome.

The Johns Hopkins Center for Bariatric Surgery (JHCBS) is designated as a Center of Excellence by the American College of Surgeons. To comply with this designation, the center must maintain a certain standard of care (SoC) and minimize complication rates. Given the potential relationship between VitD status and adverse surgical outcomes, the investigators are currently reviewing pre-operative VitD status (serum 25(OH)D concentration) collected as routine SoC and investigating the relationship with surgical outcomes under an Institutional Review Board (IRB) approved protocol (NA_00087502). The investigators findings reveal that most of bariatric surgery patients are VitD insufficient and deficient pre-operatively. To date, there is no standard regarding treating these deficiencies pre-operatively and as such the center does not intervene prior to surgery. A randomized, double-blinded, placebo-controlled pilot trial is needed to assess the causality of the relationship between pre-operative VitD status and adverse surgical outcomes in the bariatric surgical patient.

The investigators plan to identify new patients approved for bariatric surgery at the JHCBS. These patients will be randomized consecutively in a 1:1 ratio to either 30 days of 10,000 International Units (IU) of VitD3 plus SoC or 30 days of placebo plus SoC immediately prior to surgery. The investigators will monitor these patients for any adverse surgical outcomes, including wound infection, dehiscence, and prolonged length of hospital stay. The investigators will also monitor their long-term clinical outcomes such as malnutrition, weight loss, and resolution of comorbidities at their routine clinic care visit: 2 weeks, 6 weeks, 3 months, 6 months, and 12 months post-operatively. At these visits the patients are assessed for wound healing, weight loss, nutritional status, and other key markers of health, such as vital signs.

The investigators aim to determine if 10,000 IU of VitD3 daily for 30 days prior to bariatric surgery (Roux-en Y Gastric Bypass (RYGB) or Vertical Sleeve Gastrectomy (VSG)) will significantly increase the VitD status (serum 25(OH)D concentration) and whether the associated change in VitD status leads to decrease risk of adverse surgical outcomes and/or improved clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients approved for and undergoing clinically indicated bariatric surgery -Roux-en-Y Gastric Bypass (RYGBP) or Vertical Sleeve Gastrectomy (VSG)
* 18 to 64 years of age
* BMI of 35 to 49.9 kg/m2
* VitD insufficient pre-operatively: serum 25(OH)D concentration < 75 nmol/L or 30 ng/ml

Exclusion Criteria:

* Any patient who does not want to participate in the study
* Any patient who has dietary restrictions/proscriptions prohibiting ingestion of beef gelatin
* Expected poor compliance with the medical regimen
* Any active medical conditions that could, in the opinion of the investigators, jeopardize the safety of the subject or the integrity of the study
* The elective bariatric surgery is cancelled prior to incision by a surgeon for any reason
* Pregnancy: The routine standard of care is to determine whether a female patient is pregnant either by history and/or urinary pregnancy test on the day of surgery. No additional testing specifically for this study is planned beyond the standard of care.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Vitamin D status as measured by serum 25(OH)D concentration. | Up to 12 months after surgery
  Improved post-operative vitamin D status as measured by serum 25(OH)D concentration.

SECONDARY OUTCOMES:
Adverse surgical outcomes (aggregate) | Up to 30 days after surgery
  Adverse surgical outcomes include surgical site infection, wound separation and dehiscence, anastomotic leak, prolonged length of hospital stay (> 3 days), and re-admittance to the hospital within 30 days post-operatively.
Clinical outcomes (aggregate) | Up to 12 months after surgery
  Long-term clinical outcomes include wound healing, weight loss, nutritional status, resolution of comorbidities, and other key markers of health, such as vital signs (fever, blood pressure, heart rate, pain, etc.) and return of a regular menstrual cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberley E Steele, MD, PhD, Principal Investigator — Johns Hopkins University; Michael A. Schweitzer, MD, Study Director — Johns Hopkins University; Thomas H Magnuson, MD, Study Director — Johns Hopkins University
Locations (1):
- The Johns Hopkins Center for Bariatric Surgery, Baltimore, Maryland, United States

REFERENCES:
- [Background] Quraishi SA, Bittner EA, Blum L, Hutter MM, Camargo CA Jr. Association between preoperative 25-hydroxyvitamin D level and hospital-acquired infections following Roux-en-Y gastric bypass surgery. JAMA Surg. 2014 Feb;149(2):112-8. doi: 10.1001/jamasurg.2013.3176. PMID 24284777
- [Background] Goldner WS, Stoner JA, Lyden E, Thompson J, Taylor K, Larson L, Erickson J, McBride C. Finding the optimal dose of vitamin D following Roux-en-Y gastric bypass: a prospective, randomized pilot clinical trial. Obes Surg. 2009 Feb;19(2):173-179. doi: 10.1007/s11695-008-9680-y. Epub 2008 Sep 16. PMID 18795378
- [Background] Lin E, Armstrong-Moore D, Liang Z, Sweeney JF, Torres WE, Ziegler TR, Tangpricha V, Gletsu-Miller N. Contribution of adipose tissue to plasma 25-hydroxyvitamin D concentrations during weight loss following gastric bypass surgery. Obesity (Silver Spring). 2011 Mar;19(3):588-94. doi: 10.1038/oby.2010.239. Epub 2010 Oct 14. PMID 20948527
- [Background] Nguyen S, Baggerly L, French C, Heaney RP, Gorham ED, Garland CF. 25-Hydroxyvitamin D in the range of 20 to 100 ng/mL and incidence of kidney stones. Am J Public Health. 2014 Sep;104(9):1783-7. doi: 10.2105/AJPH.2013.301368. Epub 2013 Oct 17. PMID 24134366
- See also: The Johns Hopkins Center for Bariatric Surgery — http://www.hopkinsmedicine.org/johns_hopkins_bayview/medical_services/specialty_care/bariatrics/